CLINICAL TRIAL: NCT01754948
Title: Biological Monitoring of Nano Sized Particles in the Airways of Asthmatic Children
Acronym: EHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0488
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
Keywords: asthma; reactive airway disease; cough; air pollution; nano particles
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Cough

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background Ambient airborne particulate material (PM) is defined according the aerodynamic diameter into coarse, fine, and ultrafine or "nano" sized particles ranging between 2.5-10 µm (coarse), <2.5 µm (fine), and <0.1 µm (nano(. Many studies have examined particle effect on respiratory health in children, mainly by environmental monitoring of coarse and fine particles. Biological assessment of individual exposure to nano sized particles in correlation to adverse health effect was not previously studied.

Hypothesis individual exposure to nano sized particles in children is associated with reduction in forced expiratory volume at one second.

ELIGIBILITY:
Inclusion Criteria:

* age 6-18 years
* living in the Tel Aviv area
* referred to the pulmonology lab for respiratory function evaluation

Exclusion Criteria:

* Exposure to cigarette smoke
* Respiratory infection in the 4 weeks prior to recruitment and testing

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: asthmatic and control children
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
spirometry values | 1 sec
  forced expiratory volume at one second

SECONDARY OUTCOMES:
methacholine and adenosine challenge test results | 1 sec
  provocative concentration causing a 20% fall in forced expiratory volume at one second and provocative dose causing a 20% fall in forced expiratory volume at one second

CONTACTS AND LOCATIONS:
Overall Officials: Shira Benor, MD, Study Director — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel